CLINICAL TRIAL: NCT04267562
Title: Minitouch Endometrial Ablation System Treatment for Menorrhagia: An Evaluation of Safety & Effectiveness (EASE Clinical Trial)
Brief Title: Minitouch Endometrial Ablation System Treatment for Menorrhagia: An Evaluation of Safety & Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroCube, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD18036
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Menorrhagia; Heavy Menstrual Bleeding; Heavy Uterine Bleeding
Keywords: excessive menstrual bleeding; menorrhagia; heavy menstrual bleeding; heavy uterine bleeding; menstrual disorders; menstruation disturbances
MeSH Terms: conditions — Menorrhagia; Menstruation Disturbances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single-Arm, Open-Label Treatment with the Minitouch System (Other): Eligible participants will undergo a single treatment (endometrial ablation) with the Minitouch System
  Interventions: Device: Minitouch System

INTERVENTIONS:
Device: Minitouch System — The investigational treatment (endometrial ablation) will be performed utilizing the Minitouch System

SUMMARY:
The EASE Clinical Trial is prospective, multi-center, single-arm (open-label), non-randomized, clinical trial to evaluate the Minitouch Endometrial Ablation System ("Minitouch System") in premenopausal women with menorrhagia.

DETAILED DESCRIPTION:
The EASE Clinical Trial a prospective, multi-center, single-arm (open-label), non-randomized, clinical trial of the safety and effectiveness of endometrial ablation with the Minitouch System versus the FDA identified objective performance criteria (OPC) for global endometrial ablation (GEA) devices. The goal of the trial is to support reasonable safety and effectiveness of the investigational product compared to currently FDA-approved GEA devices.

Only eligible participants will undergo the Minitouch procedure. Post-treatment follow-up occurs approximately 24-hours post-procedure (via phone call) and in-person office visits occur 2-weeks, 3, 6 and 12-months post-procedure. Additional longer term follow-ups occur (via phone call or in-person office visits) 24 and 36-months post-procedure. The expected length of participation is approximately 37 months (inclusive of one month for screening and 36-months of post-procedure follow-up).

ELIGIBILITY:
Key Inclusion Criteria: Qualified participants must meet all of the following inclusion criteria.

1. Female age 30 to 50 years
2. Excessive menstrual bleeding due to benign causes
3. Uterine sounding depth measurement of 6.0 - 12.0 cm
4. A minimum uterine cavity length of 4.0 cm
5. A minimum PBLAC score of ≥ 150 for 1 menstrual cycle (obtained during screening) and must also have a documented history of excessive menstrual bleeding prior to study enrollment
6. Endometrial biopsy within 12 months prior to treatment procedure with no abnormal pathology
7. Premenopausal at screening as determined by FSH measurement ≤ 40 IU/L when age is ≥ 40 years
8. Patient agrees to use a reliable form of contraception during the study and to follow these requirements: (a) If a hormonal birth control method is used for contraception, the patient must have been on said method for ≥ 3 months prior to the onset of the screening menstrual cycle and agrees to remain on the same hormonal regimen through the initial 12-month post-treatment follow-up (pills, injections, patches, rings, implants); (b) Patient also agrees to not use hormonal birth control during the first 12-month post-treatment follow-up period if they were not using hormonal birth control during the 3 months prior to treatment
9. Ability to provide written informed consent
10. Patient is literate and clearly demonstrates understanding on how to use PBLAC after training
11. Patient agrees to the following during the study: (a) No initiation of hormonal contraception or any other medical intervention for bleeding; (b) Attend all follow-up exams through the 36-month follow-up timepoint; and (c) Exclusive use of study-provided sanitary products and submission of completed PBLAC diaries through the 12-month post-treatment follow-up

Key Exclusion Criteria: Qualified participants must NOT meet any of the following exclusion criteria.

1. Pregnant, or desires to retain fertility
2. Current or documented history of endometrial hyperplasia
3. Active endometritis
4. Clinically significant or suspected adenomyosis indicated by patient complaints, imaging, or clinician's judgment
5. Active infection of the genitals, vagina, cervix, uterus, adnexa, or urinary tract
6. Active pelvic inflammatory disease
7. Currently using an intrauterine device (IUD), including Mirena™ device, and unwilling to remove the IUD
8. Presence of an implantable contraceptive device (e.g., Essure®) protruding into the uterine cavity
9. Active sexually transmitted disease (STD) at the time of ablation
10. Presence of bacteremia, sepsis, or other active systemic infection
11. Currently on anticoagulants
12. Known clotting defects or bleeding disorders
13. Currently on medications that could thin the myometrium, such as long-term steroid use
14. Previous medical/surgical treatments, or has other conditions, that could lead to anatomic/pathologic weakness or thinning of the myometrium
15. Any general health, mental health or social situation which, in the opinion of the investigator, could represent an increased risk for the patient, or the ability of the patient to complete study requirements
16. Known/suspected abnormal uterine/pelvic anatomy or condition, such as frozen pelvis
17. Abdominal, pelvic or gynecological malignancy
18. Untreated/unevaluated cervical dysplasia, except cervical intrepithelial neoplasia I (CIN I)
19. Previous endometrial ablation procedure
20. Abnormal or obstructed, or perforated cavity as determined by investigator via standard clinical practices (e.g., hysteroscopy, saline infusion sonohysterography).
21. Intramural or subserosal myomas > 3 cm in size, or any myoma that distorts the uterine cavity
22. Any patient who is currently participating or considering participation in any other research of an investigational drug or device

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Enrollment is gender-based and is limited to females with a documented history of menorrhagia
Enrollment: 219 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott G Chudnoff, MD, MSc, Principal Investigator — Maimonides Medical Center; Amy Brenner, MD, Principal Investigator — Amy Brenner, MD & Associates, LLC
Locations (5):
- United States (5):
  - CMB Research, Newburgh, Indiana
  - Amy Brenner, MD & Associates, Mason, Ohio
  - Women's Health Texas (Women Partners in Health), Austin, Texas
  - AA ObGyn, Austin, Texas
  - OBGYN North, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 219 subjects were screened for the Trial, and 114 subjects were considered treated-enrolled. The remaining 105 subjects were excluded prior to treatment assignment for the following reasons:
  1. Trial enrollment reached: 21.9% (23/105)
  2. Withdrawn consent: 8.6% (9/105)
  3. Site closure: 5.7% (6/105)
  4. Lost to follow-up: 1.9% (2/105)
  5. Physician decision: 1.0% (1/105)
  6. Screen failure (met one or more exclusion criterion(ia)): 61.0% (64/105)
Period: Assessed for Eligibility
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 219
Completed | 114
Not Completed | 105
Not completed — Screen Failure | 64
Not completed — Trial enrollment reached | 23
Not completed — Withdrawal by Subject | 9
Not completed — Site closure | 6
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Period: Treated-Enrolled
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 114
Completed | 114
Not Completed | 0
Period: 24-Hour Contact
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 114
Completed | 114
Not Completed | 0
Period: Week 2
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 114
Completed | 114
Not Completed | 0
Period: Month 3
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 114
Completed | 114
Not Completed | 0
Period: Month 6
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 114
Completed | 114
Not Completed | 0
Period: Month 12
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 114
Completed | 114
Not Completed | 0
Period: Month 24
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 114
Completed | 112
Not Completed | 2
Not completed — Elective hysterectomy | 1
Not completed — Lost to Follow-up | 1
Period: Month 36
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Started | 112
Completed | 107
Not Completed | 5
Not completed — Elective hysterectomy | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Baseline demographics and characteristics reported for ITT Analysis Cohort.
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is calculated at day of procedure.
  years | 41.8 (4.66)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Premenopausal females | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Subjects could report more than one race, however, this is not reflected in the table due to limitations in reporting functionality.
  Participants
    American Indian or Alaska Native | 0
    Asian | 2
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 108
    More than one race | 1
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114
Baseline PBLAC (Pictorial Blood Loss Assessment Chart) Score [Mean (Standard Deviation); unit: score] — Scale information for PBLAC (Pictorial Blood Loss Assessment Chart) Score:
  The scale minimum is 0, which indicates amenorrhea, i.e., no bleeding. There is no scale maximum. A score of 100 indicates eumenorrhea, i.e., normal menstrual bleeding. A lower PBLAC score indicates less bleeding; a higher PBLAC score indicates more bleeding.
  score | 264.9 (161.39)

OUTCOME MEASURES:

1. Primary Outcome: Number of Trial Participants With Reduction in Menstrual Bleeding (PBLAC Score of ≤75)
Description: The primary effectiveness endpoint is a clinical change in menstrual blood loss as assessed by the Pictorial Blood Loss Assessment Chart (PBLAC) data, a validated, patient self-reported menstrual diary scoring system. Success for the primary effectiveness endpoint was defined as reduction in menstrual bleeding to a PBLAC (Pictorial Blood Loss Assessment Chart) score of ≤75.
  Scale information for PBLAC (Pictorial Blood Loss Assessment Chart):
  The scale minimum is 0, which indicates amenorrhea, i.e., no bleeding. There is no scale maximum. A score of 100 indicates eumenorrhea, i.e., normal menstrual bleeding. A lower PBLAC score indicates less bleeding and a higher PBLAC score indicates more bleeding.
Time Frame: Month 12 post-procedure
Population: The Intent-to-Treat (ITT) Analysis Cohort is comprised of all subjects who met all Trial eligibility criteria and in whom the procedure was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants | 102

2. Primary Outcome: Number of Trial Participants With Device or Procedure-related Serious Adverse Events
Description: The primary safety endpoint is the incidence of device or procedure-related serious adverse events.
Time Frame: Month 12 post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants | 0

3. Secondary Outcome: Number of Trial Participants That Underwent Subsequent Medical or Surgical Intervention to Treat Abnormal Bleeding
Description: Secondary safety outcome measures are the number of trial participants that underwent medical or surgical intervention to treat abnormal bleeding.
Time Frame: Month 12 post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants | 0

4. Secondary Outcome: Number of Trial Participants That Underwent Subsequent Medical or Surgical Intervention to Treat Abnormal Bleeding
Description: as for outcome 3
Time Frame: >Month 12 through Month 24 post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 112
Participants | 2

5. Secondary Outcome: Number of Trial Participants That Underwent Subsequent Medical or Surgical Intervention to Treat Abnormal Bleeding
Description: as for outcome 3
Time Frame: >Month 24 through Month 36 post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants | 1

6. Secondary Outcome: Number of Trial Participants With Amenorrhea
Description: Secondary Effectiveness Outcome Measure - Amenorrhea rates where PBLAC = 0 (no bleeding)
Time Frame: Month 6 and Month 12 post-procedure
Population: The Per Protocol (PP) Analysis Cohort is comprised of all Intent-to-Treat (ITT) subjects who are treatable, completed the ablation procedure, and attended the 12-month follow-up visit.
Measure: Number; unit: participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
participants
  Month 6 | 50
  Month 12 | 59

7. Secondary Outcome: Number of Trial Participants With Amenorrhea
Description: Secondary Effectiveness Outcome Measure - Amenorrhea rates per the Investigator Global Evaluation (IGE)
Time Frame: Month 24 post-procedure
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 112
participants | 49

8. Secondary Outcome: Number of Trial Participants With Amenorrhea
Description: Secondary Effectiveness Outcome Measure - Amenorrhea rates per the Investigator Global Evaluation (IGE)
Time Frame: Month 36 post-procedure
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 107
participants | 48

9. Secondary Outcome: Dysmenorrhea-related Pain Score
Description: Change in quality of life as measured by Dysmenorrhea-related pain score using the Numerical Rating Scale (NRS) (scale of minimum 0 to maximum 10, where 0 = no pain, 5 = moderate pain, 10 = worst pain). A higher score indicates a worse outcome.
Time Frame: Baseline, Month 6 and Month 12 post-procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
score on a scale
  Baseline | 6.1 (2.6)
  Month 6 | 0.9 (1.5)
  Month 12 | 0.8 (1.5)

10. Secondary Outcome: Dysmenorrhea-related Pain Score
Description: as for outcome 9
Time Frame: Baseline and Month 24 post-procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 112
score on a scale
  Baseline | 6.2 (2.6)
  Month 24 | 1.0 (1.8)

11. Secondary Outcome: Dysmenorrhea-related Pain Score
Description: as for outcome 9
Time Frame: Baseline and Month 36 post-procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 107
score on a scale
  Baseline | 6.2 (2.6)
  Month 36 | 0.9 (1.7)

12. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 2) - Limitations in Work Outside or Inside the Home
Description: Change in quality of life as measured by Menorrhagia Impact Questionnaire (MIQ 2):
  Subjects were asked if they had any limitations in work outside or inside the home based on the following categories: not at all, slightly, moderately, quite a bit, extremely
Time Frame: Baseline, Month 6 and Month 12 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants
  Baseline: Not at all | 9
  Baseline: Slightly | 17
  Baseline: Moderately | 34
  Baseline: Quite a bit | 34
  Baseline: Extremely | 20
  Month 6: Not at all | 105
  Month 6: Slightly | 7
  Month 6: Moderately | 2
  Month 6: Quite a bit | 0
  Month 6: Extremely | 0
  Month 12: Not at all | 108
  Month 12: Slightly | 3
  Month 12: Moderately | 3
  Month 12: Quite a bit | 0
  Month 12: Extremely | 0

13. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 2) - Limitations in Work Outside or Inside the Home
Description: as for outcome 12
Time Frame: Baseline and Month 24 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 112
Participants
  Baseline: Not at all | 9
  Baseline: Slightly | 17
  Baseline: Moderately | 33
  Baseline: Quite a bit | 33
  Baseline: Extremely | 20
  Month 24: Not at all | 101
  Month 24: Slightly | 7
  Month 24: Moderately | 1
  Month 24: Quite a bit | 3
  Month 24: Extremely | 0

14. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 2) - Limitations in Work Outside or Inside the Home
Description: as for outcome 12
Time Frame: Baseline and Month 36 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 107
Participants
  Baseline: Not at all | 8
  Baseline: Slightly | 15
  Baseline: Moderately | 32
  Baseline: Quite a bit | 32
  Baseline: Extremely | 20
  Month 36: Not at all | 100
  Month 36: Slightly | 5
  Month 36: Moderately | 1
  Month 36: Quite a bit | 1
  Month 36: Extremely | 0

15. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 3) - Limitations in Physical Activity
Description: Change in quality of life as measured by Menorrhagia Impact Questionnaire (MIQ 3):
  Subjects were asked if they had any limitations in physical activity based on the following categories: not at all, slightly, moderately, quite a bit, extremelylimitations in social and leisure activities: not at all, slightly, moderately, quite a bit, extremely
Time Frame: Baseline, Month 6 and Month 12 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants
  Baseline: Not at all | 2
  Baseline: Slightly | 20
  Baseline: Moderately | 27
  Baseline: Quite a bit | 40
  Baseline: Extremely | 25
  Month 6: Not at all | 107
  Month 6: Slightly | 6
  Month 6: Moderately | 1
  Month 6: Quite a bit | 0
  Month 6: Extremely | 0
  Month12: Not at all | 106
  Month12: Slightly | 5
  Month12: Moderately | 2
  Month12: Quite a bit | 1
  Month12: Extremely | 0

16. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 3) - Limitations in Physical Activity
Description: as for outcome 15
Time Frame: Baseline and Month 24 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 112
Participants
  Baseline: Not at all | 2
  Baseline: Slightly | 20
  Baseline: Moderately | 27
  Baseline: Quite a bit | 38
  Baseline: Extremely | 25
  Month 24: Not at all | 98
  Month 24: Slightly | 10
  Month 24: Moderately | 1
  Month 24: Quite a bit | 3
  Month 24: Extremely | 0

17. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 3) - Limitations in Physical Activity
Description: as for outcome 15
Time Frame: Baseline and Month 36 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 107
Participants
  Baseline: Not at all | 1
  Baseline: Slightly | 19
  Baseline: Moderately | 25
  Baseline: Quite a bit | 37
  Baseline: Extremely | 25
  Month 36: Not at all | 100
  Month 36: Slightly | 4
  Month 36: Moderately | 2
  Month 36: Quite a bit | 1
  Month 36: Extremely | 0

18. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 4) - Limitations in Social or Leisure Activities
Description: Change in quality of life as measured by Menorrhagia Impact Questionnaire (MIQ 4):
  Subjects were asked if they had any limitations in social or leisure activities based on the following categories: not at all, slightly, moderately, quite a bit, extremely
Time Frame: Baseline, Month 6 and Month 12 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants
  Baseline: Not at all | 7
  Baseline: Slightly | 20
  Baseline: Moderately | 30
  Baseline: Quite a bit | 36
  Baseline: Extremely | 21
  Month 6: Not at all | 107
  Month 6: Slightly | 6
  Month 6: Moderately | 1
  Month 6: Quite a bit | 0
  Month 6: Extremely | 0
  Month 12: Not at all | 108
  Month 12: Slightly | 4
  Month 12: Moderately | 1
  Month 12: Quite a bit | 1
  Month 12: Extremely | 0

19. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 4) - Limitations in Social or Leisure Activities
Description: as for outcome 18
Time Frame: Baseline and Month 24 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 112
Participants
  Baseline: Not at all | 7
  Baseline: Slightly | 20
  Baseline: Moderately | 28
  Baseline: Quite a bit | 36
  Baseline: Extremely | 21
  Month 24: Not at all | 101
  Month 24: Slightly | 7
  Month 24: Moderately | 2
  Month 24: Quite a bit | 1
  Month 24: Extremely | 1

20. Secondary Outcome: Menorrhagia Impact Questionnaire (MIQ 4) - Limitations in Social or Leisure Activities
Description: as for outcome 18
Time Frame: Baseline and Month 36 post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 107
Participants
  Baseline: Not at all | 6
  Baseline: Slightly | 19
  Baseline: Moderately | 26
  Baseline: Quite a bit | 36
  Baseline: Extremely | 20
  Month 36: Not at all | 102
  Month 36: Slightly | 3
  Month 36: Moderately | 1
  Month 36: Quite a bit | 1
  Month 36: Extremely | 0

21. Secondary Outcome: Procedure Details: Number of Trial Participants in Which a Cervical Dilator Was Used
Description: Secondary Outcome Measure - Use of Cervical Dilator (Yes / No) Time frame: the need for using a cervical dilator is assessed on day of procedure, during the procedure
Time Frame: Day of Procedure (during the procedure)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants
  Yes - cervical dilator used | 9
  No - cervical dilator not used | 105

22. Secondary Outcome: Procedure Details: Type of Setting in Which the Procedure Took Place
Description: Secondary Outcome Measure - Setting in which the Minitouch Procedure took place Time frame: the type of setting is assessed on day of procedure, prior to the procedure
Time Frame: Day of Procedure (prior to the procedure)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants
  Physician's office | 114
  Outpatient clinic/facility (surgery center) | 0
  Affiliated hospital | 0

23. Secondary Outcome: Procedure-related Pain Score
Description: Procedure-related pain score using the Numerical Rating Scale (NRS) (scale of minimum 0 to maximum 10, where 0 = no pain, 5 = moderate pain, 10 = worst pain). A higher score indicates a worse outcome.
  Timepoints:
  Pre-procedure (on the day of, prior to the procedure) Discharge (post-procedure, prior to discharge) 24-hours post-procedure (18-48 hours post-procedure)
Time Frame: Pre-Procedure (on day of, prior to procedure), Discharge (post-procedure, prior to discharge) and 24-hours post-procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
score on a scale
  Pre-procedure (on the day of, prior to the procedure | 0.6 (1.5)
  Discharge (post-procedure, prior to discharge) | 2.6 (2.4)
  24-hours post-procedure (18-48 hours post-procedure) | 1.2 (1.5)

24. Secondary Outcome: Procedure Details: Recovery Time
Description: Secondary Outcome Measure - Total Procedure Recovery Time Time frame: assessed on the day of procedure/post-procedure, prior to discharge
Time Frame: Day of Procedure (post-procedure, prior to discharge)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
minutes | 20.8 (22.7)

25. Other Pre Specified Outcome: Additonal Measure - Subject Self-Report of Pregnancy
Description: Count of subject self-report of pregnancy at Month 36 to satisfy the post-approval study (PAS) reporting requirements
Time Frame: Month 36 post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 107
Participants | 0

26. Other Pre Specified Outcome: Additonal Measure - Contraception Status at Month 36
Description: Count of subject contraception menthods reported at Month 36 to satisfy the post-approval study (PAS) reporting requirements; subjects could report more than one method of contraception so numbers may be greater than the total of subjects
Time Frame: Month 36 post-procedure
Measure: Number; unit: participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 107
participants
  Abstinence | 5
  Condom | 21
  Partner's vasectomy | 48
  Tubal sterilization | 30
  Hormonal method (includes pills, injections, rings, implants) | 4
  Intrauterine devices | 2
  Other (includes no method of contraception) | 4

27. Other Pre Specified Outcome: Additonal Measure - Gynecologic Adverse Events
Description: Count of number of subjects that reported gynecologic adverse events through Month 24 and Month 36;
Time Frame: Month 24 and Month 36 post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
Number analyzed (Participants) | 114
Participants
  >Month 12 to Month 24: Bacterial vaginosis | 1
  >Month 12 to Month 24: Urinary tract infection | 4
  >Month 12 to Month 24: Bladder pain | 1
  >Month 12 to Month 24: Renal colic | 1
  >Month 12 to Month 24: Renal mass | 1
  >Month 12 to Month 24: Stress urinary incontinence | 1
  >Month 12 to Month 24: Ureterolithiasis | 1
  >Month 12 to Month 24: Urinary incontinence | 1
  >Month 12 to Month 24: Anxiety | 1
  >Month 12 to Month 24: Coital bleeding | 1
  >Month 12 to Month 24: Menopausal symptoms | 1
  >Month 12 to Month 24: Ovarian cyst | 1
  >Month 12 to Month 24: Uterine hemorrage | 1
  >Month 24 to Month 36: Bacterial vaginosis | 1
  >Month 24 to Month 36: Urinary tract infection | 1
  >Month 24 to Month 36: Dysuria | 1
  >Month 24 to Month 36: Dysmenorrhea | 2
  >Month 24 to Month 36: Ovarian cyst | 1

ADVERSE EVENTS:
Time Frame: Month 36 post-procedure
Description: The protocol defines an adverse event (AE) as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the medical device. This includes any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medical device, whether or not related to the medical device. Therefore, all adverse events regardless of causality are reported.
Arm/Group | Single-Arm, Open-Label Treatment With the Minitouch System
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 3/114
Other Adverse Events (participants affected / at risk) | 109/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Arm, Open-Label Treatment With the Minitouch System (N=114)
Atrial fibrillation (Cardiac disorders) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Arm, Open-Label Treatment With the Minitouch System (N=114)
Postural orthostatic tachycardia syndrome (POTS) (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Eustachian tube disorder (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Blindness (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Procedural nausea (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Hypensensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 33 (33)
Cellulitis (Infections and infestations) | 1 (1)
Cholera (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Pharyngitis streptoccal (Infections and infestations) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (7)
Vaginal infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Arthropod sling (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Blood testosterone decreased (Investigations) | 1 (1)
Mammogram abnormal (Investigations) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Glucose intolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Restless leg syndrome (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1) — not related to the investigational device
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (7)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 2 (2)
Stress (Psychiatric disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Coital bleeding (Reproductive system and breast disorders) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (3)
Stress urinary incontinence (Reproductive system and breast disorders) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 2 (2)
Uterine spasm (Reproductive system and breast disorders) | 50 (50)
Vaginal discharge (Reproductive system and breast disorders) | 4 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal odour (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Autoimmune dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Menopause (Social circumstances) | 1 (1)
Medical device change (Surgical and medical procedures) | 1 (1)
Hot flush (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Bacterial vaginosis (Infections and infestations) | 6 (6)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Abdominal pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 5 (5)
Near syncope (vasovagal response) (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04267562/Prot_SAP_000.pdf